CLINICAL TRIAL: NCT01408199
Title: Phase II Study To Evaluate The Safety And Efficacy Of Lenalidomide For The Treatment Of Refractory Cutaneous Lupus
Brief Title: Study To Evaluate The Safety And Efficacy Of Lenalidomide For Refractory Cutaneous Lupus
Acronym: ORDI-02
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: RESEARCH INSTITUTE, VALL D'HEBRON HOSPITAL
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-016508-21
Record Dates: First submitted 2011-07-19; First posted 2011-08-03 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2011-08

CONDITIONS: Cutaneous Lupus
Keywords: Lenalidomide; Refractory Cutaneous Lupus
MeSH Terms: interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide Group (Experimental)
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — 5 mg daily will be administered until the achievement of complete response, and then tapered progressively according to clinical response

SUMMARY:
Cutaneous Lupus is frequent. Approximately 70% of patients with SLE will develop cutaneous involvement at some point during course of their disease. In spite of the esthetic consequence during the acute phase, the main problem is still related to its disfiguring and incapacitating nature. Topical steroids and/or antimalarial therapy continue to be the conventional therapy. Unfortunately, approximately 30% will be refractory to these measures. For those patients, immunosuppressive therapy can be an alternative with controversial results. Several series have shown a 90% of clinical efficacy in patients treated with Thalidomide. Unfortunately, the main drawback has been the serious described side effects such as fetal malformations, polyneuropathy and drowsiness. Recently, a new thalidomide analogue, more potent, efficient and with better safety profile has been discovered. The main objective of the study is to evaluate the efficacy and safety of Lenalidomide for patients with Refractory cutaneous Lupus. Secondary objectives include evaluating the effect of this drug on the systemic manifestations of lupus disease, the adverse effects, frequency of flare after withdrawal, the sequela and the effect on the seric parameters. Methods: Twelve patients with refractory cutaneous lupus will be included. Lenalidomide will be started at 5mg/day and tapered progressively. Blood test and EMG will be performed at onset and at the end of follow up.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Histologically proven cutaneous lupus erythematosus with or without associated systemic disease
* Presence of at least a grade II erythema as assessed by the validated modified Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI)
* Cutaneous lesions involving more than 18% of the body surface calculated according to the rule of the nines, or history of severe side effects or lack of efficacy following thalidomide therapy, in cutaneous lupus disease refractory to conventional treatment with antimalarials and topical steroids.
* No pregnancy or wish to become pregnant during the study period.

Exclusion Criteria:

* Pregnancy, breastfeeding or the use of not adequate contraception.
* Severe thrombocytopenia (<30x10E9 cells/L) or leucopoenia (<1500x10E9), known at least 30 days prior to the onset of the study,
* Previous history of arterial/venous thrombosis,
* Presence of antiphospholipid antibodies
* Presence of moderate-severe renal impairment (FG <30 ml/min)
* Progressive renal disease.
* Lack of written informed consent prior to participation in the study.
* Presence of a concomitant systemic flare that may require other systemic treatments for its control
* Any psychiatric o social disease that may interfere with the study and follow-up
* HIV, B or C hepatitis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-01; Primary Completion 2010-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving a complete response | 3 months
  Clinical response will be evaluated by the validated CLASI score. Complete response will be considered when CLASI score=0 following treatment.
Proportion of patients developing a side effect | 12 months

SECONDARY OUTCOMES:
Proportion of patients developing a systemic lupus flare | 6 months
  Systemic activity will be assess by the SLEDAI score. Disease activity will be considered with a SLEDAI score > or = 6.
Proportion of patients increasing anti-dsDNA levels | 12 months
  Anti-dsDNA titers will be mesured by ELISA at each visist.
Proportion of patients having a cutaenous flare following treatment withdrawal | 12 months
  Cutaneous flare will be defined by at least one CLASi > or= 2 in those patients with a previous complete resolution of the inflammatory rash (CLASI=0)
Proportion of patients with an increase CLASI damage score following treatment. | 12 months
  Sequelae will be evaluated but the CLASI score, damage area. Any increase in the score compared to initial scores will be considered as sequelae.

CONTACTS AND LOCATIONS:
Overall Officials: JOSEP ORDI-ROS, M, Principal Investigator — VALL D'HEBRON HOSPITAL
Locations (1):
- Vall D'Hebron Hospital, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Cortes-Hernandez J, Avila G, Vilardell-Tarres M, Ordi-Ros J. Efficacy and safety of lenalidomide for refractory cutaneous lupus erythematosus. Arthritis Res Ther. 2012 Dec 7;14(6):R265. doi: 10.1186/ar4111. PMID 23217273